CLINICAL TRIAL: NCT03836235
Title: Development of a Risk Prediction Screening Tool for Opioid-Prescription Injury (STOP Injury) in Older Adults Initiated on Opioids From the Emergency Department
Acronym: STOP Injury
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB201802137- N; R33AG056540 (NIH); JAX ASCENT Junior Scholar (Other Grant/Funding Number: US Department of Health and Human Services)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Opioid Use
Keywords: older adults; quality of life; adverse events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mouthwash samples will be used to test for the presence of single-nucleotide polymorphisms (CYP2D6, OPRM1, COMT, ABCB1, OCT1) in the genes that mediate opioid metabolism.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The long-term goal of this project is to promote responsible opioid prescribing, immediately improving patient safety and ultimately decreasing healthcare costs by reducing older adult morbidity and mortality due to opioid-related injury. The objective of this pilot project is to gather data to inform the development of the STOP Injury tool and evaluate additional predictive factors and important outcomes relevant to prescription opioids.

DETAILED DESCRIPTION:
The experience from this project will lay the groundwork on prospective validation of STOP Injury in a large appropriately powered study. Aim 1 will provide data that will help narrow inclusion of candidate variables in the STOP Injury tool to include those that are most feasible to collect and most predictive. Aim 2 will help inform the possible inclusion of genetic factors into a predictive model. Finally, Aim 3 will help identify quality of life outcomes that should be considered when assessing opioid medication adverse events.

Aim 1. Evaluate the association between prescription opioid adverse events in older adults and candidate risk prediction variables proposed for STOP Injury prediction score The study team will conduct a pilot prospective observational study of 200 patients 50 years or older who are initiated on opioids from the emergency department (ED). The investigators will analyze the association between candidate risk factors and opioid adverse events (falls and OD).

Aim 2. Evaluate the association between prescription opioid adverse events and genetic factors.

In the cohort from Aim 1, the study team will test subjects for 12 genetic single nucleotide polymorphisms related to opioid metabolism, transport, and effect.

Aim 3. Measure the impact of opioid medications on quality of life measures in older adults The investigators will implement a series of quality of life measures on a subset of patients as a pilot study to determine which measures capture the impact prescription opioids have on older adults' quality of life

ELIGIBILITY:
Inclusion Criteria:

* Presenting to UF JAX ED with pain or a pain-related complaint (i.e., fracture, burn, etc.)
* Patient has not used opioids 15 days or more within the last 30 days
* Patient does not have opioid medications at home
* Discharge to home with an opioid prescription

Exclusion Criteria:

* Bed-bound or uses wheelchair
* Living in skilled nursing facility or assisted living facility
* Non-English speaking
* Unable to provide consent
* Incarcerated
* Lack of reliable telephone access
* Use of opioids on most days for >3 months

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will seek to enroll 200 subjects. All patients 50 years or older presenting to UF JAX ED with pain or a pain-related complaint (i.e., fracture, burn, etc.) will be screened for eligibility using the inclusion and exclusion criteria listed below. To accomplish Aim 3, the investigators will enroll a convenience subset of patients by approaching every third subject enrolled with the option to consent for Aim 3.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Safety, as measured by number of subjects with at least one fall adverse event | Up to 30 days
  The study team will analyze the association between candidate risk factors and opioid adverse events (falls and OD).

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Sheikh, MD, Principal Investigator — UF College of Medicine--Jacksonville
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No